CLINICAL TRIAL: NCT03572660
Title: Phase II Study Assessing the Combined Use of Autologous Bone Marrow Derived Mononuclear Cells and G-csf With Percutaneous Circulatory Assistance in the Treatment of Dilated Cardiomyopathy
Brief Title: Use of Bone Marrow Derived Stem Cell and G-CSF With Circulatory Assistance in the Treatment of DCM
Acronym: DCM-Support
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Reda 012357; 2018-001063-23 (EudraCT Number)
Record Dates: First submitted 2018-03-29; First posted 2018-06-28 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Dilated Cardiomyopathy
Keywords: Stem Cell; Circulatory Support; Heart Failure; G-CSF
MeSH Terms: conditions — Cardiomyopathy, Dilated; Heart Failure | interventions — Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Intervention Model Description: Single arm intervention study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BMMNC intervention arm (Other): Bone marrow derived mononuclear cells and G-CSF
  Interventions: Biological: Bone marrow derived mononuclear cells and G-CSF

INTERVENTIONS:
Biological: Bone marrow derived mononuclear cells and G-CSF — Intra-coronary infusion

SUMMARY:
DCM Support is recruiting patients with dilated cardiomyopathy and heart failure symptoms. The goal of this clinical trial is to examine whether treatment with a patient's own stem cells can improve their heart function and alleviate heart failure symptoms.

* Stem cells will be collected from bone marrow in the patient's hip under local anaesthetic.
* The stem cells will be infused into the arteries that supply blood to the heart under local anaesthetic.
* A mini heart pump will be used to take the strain off the heart during the procedure.
* The follow-up involves a phone call at 1 month and clinic visits at 3 and 12 months

DETAILED DESCRIPTION:
DCM SUPPORT is a single centre, single arm clinical trial taking place at St Bartholomew's Hospital in London, UK.

* It is recruiting patients with dilated cardiomyopathy and ongoing heart failure symptoms
* All patients undergo a bone marrow aspiration after 5 days of subcutaneous G-CSF injections
* After cell processing, bone marrow-derived mononuclear cells are infused into the coronary arteries using the stop-flow technique. An intra-procedural Impella CP device is used to support the circulation.
* The primary endpoint is change in left ventricular ejection fraction at 3 months as measured by cardiac CT.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of dilated cardiomyopathy under the supervision of a physician or a heart failure nurse specialist.
* NYHA class ≥ 2 symptoms despite having received optimal medical therapy and appropriate device therapy, as per clinical guidelines for an interval of at least 3 months.
* No other treatment options available as part of the current best standard of care.
* LVEF ≤35% on any imaging modality performed as part of the screening phase.

Exclusion Criteria:

* Congenital heart disease.
* Clinically significant valvular heart disease.
* Patients who are not suitable for a Percutaneous Mechanical Support Device (E.g. unsuitable femoral artery anatomy, unable able to lie flat for prolonged time to accommodate the stem cell infusion & presence of LV thrombus)
* Weight of patient that exceeds the maximum limit of the cardiac catheterisation laboratory table / CT scanner.
* Cardiomyopathy 2o to a reversible cause that has not been treated e.g. thyroid disease, alcohol abuse, hypophosphataemia, hypocalcaemia, cocaine abuse, selenium toxicity & chronic uncontrolled tachycardia.
* Cardiomyopathy in association with a neuromuscular disorder e.g. Duchenne's progressive muscular dystrophy.
* Previous cardiac surgery.
* Contra-indication for bone marrow aspiration (thrombocytopaenia - platelet count <80 x 10(9)/L or extensive surgical scarring/anatomical deformity at site of bone marrow puncture).
* Known active infection on admission as defined by a temperature >37.5°C or on a short course of antibiotics.
* An active infection of hepatitis B, hepatitis C, syphilis or HTLV
* Known HIV infection
* Chronic inflammatory disease requiring on-going medication.
* Concomitant disease with a life expectancy of less than one year
* Follow-up impossible (no fixed abode, etc.)
* Neoplastic disease without documented remission within the past 5 years.
* Patients on renal replacement therapy.
* Subjects of childbearing potential unless βHCG negative and are on adequate contraception during the trial.
* Patients falling into the vulnerable category or lacking capacity
* Patients who are unable to understand or read written English will be excluded from the trial.
* Killip Class III or above

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-12-24 (Actual); Primary Completion 2030-03-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in left ventricular ejection fraction | Baseline to 3 months
  Change in left ventricular ejection fraction as measured by cardiac CT

SECONDARY OUTCOMES:
Change in left ventricular ejection fraction | Baseline to 12 months
  Change in left ventricular ejection fraction as measured by cardiac CT
Change in exercise capacity | Baseline to 3 and 12 months
  Change in exercise capacity as assessed by a 6-minute walk test
Change in heart failure symptoms | Baseline to 3 and 12 months
  Change in heart failure symptoms as measured by NYHA classification
Change in quality of life as assessed by Minnesota Living with Heart Failure Questionnaire scores | Baseline to 3 and 12 months
  Change in quality of life as measured by MLHFQ (The 21-item MLHFQ uses a 6-point Likert scale, where 0 = no, 1= very little and 5= very much. The questions are intended to be representative of the ways heart failure can affect physical and emotional dimensions of quality of life)
Change in quality of life as measured by EuroQol-5 Dimension 5 Levels questionnaires | Baseline to 3 and 12 months
  Change in quality of life as measured by EQ-5D-5L questionnaires (the scale measures quality of life on a 5-component scale including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression)
Procedural safety as assessed by in-hospital procedural related morbidity/mortality | In-hospital procedural time
  Procedural safety as assessed by in-hospital procedural related morbidity/mortality
Change in biochemical markers of heart failure | Baseline to 3 and 12 months
  Change in biochemical markers of heart failure as measured by change in NT-proBNP
Assessment of rates of MACE (cumulative & individual components) | 3 and 12 months
  Rates of MACE (all-cause death, myocardial infarction, hospitalisation for heart failure, major arrhythmias [defined as VT and VF])
Assessment of rates of stroke | 3 and 12 months
  Assessment of rates of stroke
Assessment of peri-procedural myocardial infarction | Day 0 and Day 6
  Assessment of peri-procedural myocardial infarction as per SCAI definition measured by change in troponin (MI defined by increase in troponin >70 times upper limit of normal from baseline).
Change in renal function | Baseline to 3 and 12 months
  Change in renal function from baseline at 3 and 12 months as measured by creatinine levels.
Change in inflammatory markers | Baseline to 3 and 12 months
  Change in inflammatory markers as measured by change in C-reactive protein

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Mathur, Principal Investigator — Queen Mary University of London
Locations (1):
- St Bartholomew's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fawaz S, Ramaseshan R, Khan S, Davies JR, Collet C, Karamasis GV, Cook CM, Jones DA, Mathur A, Keeble TR. Left Ventricular Unloading in Nonischemic Dilated Cardiomyopathy Improves Coronary Haemodynamic Reserve. Catheter Cardiovasc Interv. 2025 Jun;105(7):1719-1722. doi: 10.1002/ccd.31514. Epub 2025 Mar 27. PMID 40145630
- [Derived] Reid A, Hussain M, Veerapen J, Ramaseshan R, Hall R, Bowles R, Jones DA, Mathur A. DCM Support: cell therapy and circulatory support for dilated cardiomyopathy patients with severe ventricular impairment. ESC Heart Fail. 2023 Aug;10(4):2664-2671. doi: 10.1002/ehf2.14393. Epub 2023 May 15. PMID 37190883